CLINICAL TRIAL: NCT03250299
Title: Phase I Study to Determine the Safety and Tolerability of the Oral Microtubule Destabilizer BAL101553 in Combination With Standard Radiation in Patients With MGMT Promoter Unmethylated Newly Diagnosed Glioblastoma
Brief Title: Microtubule-Targeted Agent BAL101553 and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the National Cancer Institute's (NCI)-mandated termination of the Adult Brain Tumor Consortium which was conducting the study
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABTC 1601; CDI-CS-004 (Other: Basilea); IRB00131687 (Other: JHM IRB)
Record Dates: First submitted 2017-07-28; First posted 2017-08-15 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma; MGMT-Unmethylated Glioblastoma
Keywords: Glioblastoma; Brain tumor; Lisavanbulin; BAL101553
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — lisavanbulin; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Finding (Experimental): Fixed 3+3 dose escalation of BAL101553 (7 days per week), combined with RT days 1-5 for 6 weeks followed by 4 week rest.
  Interventions: Drug: Microtubule-Targeted Agent BAL101553; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Microtubule-Targeted Agent BAL101553 — Given PO
  Other Names: BAL101553, Microtubule-targeted Agent BAL101553
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy, Irradiate, irradiated, irradiation, RADIATION, Radiation, radiation therapy, Radiation Therapy, Radiotherapeutics, radiotherapy, Radiotherapy, RT, Therapy, Radiation

SUMMARY:
This Phase I study investigated the side-effects and best dose of microtubule-targeted agent BAL101553 when given together with radiation therapy in treating patients with newly-diagnosed O6-methylguanine-DNA methyltransferase (MGMT) promoter unmethylated glioblastoma (GBM). Drugs used in chemotherapy, such as microtubule-targeted agent BAL101553, work in different ways to stop the growth of tumor cells, either by killing the cells, stopping them from dividing, or stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving microtubule-targeted agent BAL101553 and radiation therapy may work better in treating patients with GBM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of microtubule-targeted agent BAL101553 (BAL101553) in combination with standard radiation in patients with newly diagnosed MGMT promoter unmethylated GBM.

SECONDARY OBJECTIVES:

I. To estimate safety and tolerability of the combination of BAL101553 in combination with standard radiation in patients with newly diagnosed MGMT promoter unmethylated GBM.

II. To determine overall and progression-free survival.

OUTLINE: This was a dose escalation study of the microtubule-targeted agent BAL101553.

Patients received BAL101553 orally (PO) once daily (QD) for 6 weeks, concurrent with standard radiation therapy (RT) 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity.

This treatment period was followed by a 4-week no-treatment period. The duration of study treatment was defined as these 6 weeks of treatment plus the 4 weeks of rest.

The safety evaluation period was the 10 weeks from start of treatment

After completion of study treatment, patients were followed up at 30 days, and then every 2 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
The following inclusion criteria were applied:

* Patients must have had histologically-proven GBM
* Patients must have recovered from the immediate post-operative period
* Patients must have had tumor MGMT methylation status of unmethylated as determined by local pathologist using a Clinical Laboratory Improvement Act (CLIA)-approved diagnostic test; results of routinely-used methods for MGMT methylation testing (e.g. methylation-specific [MS]- polymerase chain reaction [PCR] or quantitative PCR) were acceptable
* Patients must have been be able to undergo magnetic resonance imaging (MRI) of the brain with gadolinium
* Patients must not have received prior radiation therapy (RT), chemotherapy, immunotherapy or therapy with a biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed
* Patients must have had a tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of GBM, completed and signed by a pathologist
* Patients must have had a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/micro liter (mcL)
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), unless the patient has known Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Creatinine =< 1.5 x ULN
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > ULN
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x ULN
* Sodium >= 130 mmol/L
* Patients must have been able to provide written informed consent
* Patients must have had baseline MRI performed within the 21 days prior to starting treatment
* Women of childbearing potential must have had a negative serum pregnancy test within 72 hours prior to the first dose of BAL101553; women of childbearing potential must have agreed to use highly-effective contraceptive methods for the duration of study participation and for an additional 90 days after the last dose of study drug; highly-effective contraceptive methods include male or female sterilization (bilateral tubal occlusion or vasectomy); intrauterine device (IUD); combined (estrogen- and progesterone-containing) hormonal contraception (oral, vaginal ring or transdermal patch) with an ethinylestradiol dose of at least 30 ug, plus use of male condoms (preferably with spermicides), female condoms, a female diaphragm or a cervical cap; or total sexual abstinence; if a woman became pregnant or suspected she was pregnant while participating in this study, she was asked to inform her treating physician immediately; male patients must have agreed not to donate sperm from the time of the first dose of study drug until 90 days after the end of treatment; male patients, without a vasectomy and with a partner of childbearing potential, must have agreed to use condoms during the study and for at least 90 days after the end of treatment; the patient should have been instructed that their female partner should use another form of contraception for the duration of the study and continue this use for at least 90 days after the last dose of study drug
* Patients must have had no concurrent malignancies except curatively-treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must have been disease-free for >= 5 years
* Patients must have been maintained on a stable corticosteroid regimen (no increase for 5 days) prior to the start of treatment
* Patients must have been able to swallow whole capsules

The following exclusion criteria were applied:

* Patients receiving any other investigational agent
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to BAL101553
* Patients on drugs that are strong inhibitors and/or inducers of CYP2C9, CYP2C19 or CYP3A4 (including enzyme-inducing anti-epileptic drugs EIAEDs]), were not eligible for the study; patients taking non-EIAEDs were permitted to take part in the study; patients previously treated with any of the prohibited concomitant medications listed above may have been enrolled if they had been off the medication for >= 10 days prior to the first dose of BAL101553
* Patients may not have been on coumarin anti-coagulants (warfarin, etc.); heparin, low-molecular weight heparin (LMWH), or other antithrombotic medications were permitted
* Patients with gastrointestinal disease, or those who had a procedure that was expected to interfere with the oral absorption or tolerance of BAL101553 (e.g., functionally-relevant gastrointestinal obstruction, or frequent vomiting unresolved upon anti-emetic supportive care)
* Patients with peripheral neuropathy >= Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Patients with ataxia >= CTCAE grade 2
* Patients with known acute or chronic hepatitis B or hepatitis C infection
* Patients with systolic blood pressure (SBP) >= 140 mmHg or diastolic blood pressure (DBP) >= 90 mmHg at the screening visit were ineligible; patients with an initial clinic blood pressure (BP) >= 140/90 mmHg may be included if SBP < 140 mmHg and DBP < 90 mmHg is confirmed in two subsequent BP measurements on the same day
* Patients with BP combination treatment with more than two antihypertensive medications were ineligible
* Significant cardiac disease or abnormality, including any of the following:

  * Left ventricular ejection fraction < 50% at screening (assessed by echocardiography, cardiac MRI or multigated acquisition [MUGA])
  * Corrected QT Fridericia's correction formula (QTcF) > 470 ms on screening electrocardiogram (ECG), or a clinically-relevant ECG abnormality
  * Congenital long QT syndrome
  * History of sustained ventricular tachycardia, ventricular fibrillation, or torsades de pointes
  * Presence of atrial fibrillation with tachyarrhythmia (ventricular response rate > 100 beats per minute [bpm])
  * Bradycardia (heart rate < 50 bpm)
  * Complete left bundle branch block.
  * Bifascicular block (complete right bundle branch block and anterior or posterior left hemiblock)
  * Myocardial infarction, acute coronary syndrome (including unstable angina), coronary revascularization procedures, or coronary arterial bypass grafting within the 6 months prior to starting study drug
  * Cardiac troponin (either troponin T or troponin I) > ULN
  * Congestive heart failure of New York Heart Association class III or IV
  * Unstable angina pectoris
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, were ineligible
* Pregnant women were excluded from this study; breastfeeding should have been discontinued if the mother was treated with BAL101553
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy were ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Holdhoff, MD, Study Chair — National Cancer Institute (NCI)
Locations (8):
- United States (8):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment was administered on an outpatient basis
Groups:
- BAL101553 4 mg Cohort: BAL101553 was given as an 4 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 6 mg Cohort: BAL101553 was given as an 6 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 8 mg Cohort: BAL101553 was given as an 8 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 12 mg Cohort: BAL101553 was given as an 12 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 15 mg Cohort: BAL101553 was given as an 15 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
Period: BAL101553 4 mg Cohort
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Started | 5 | 0 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: BAL101553 6 mg Cohort
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Started | 0 | 5 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0 | 0
Period: BAL101553 8 mg Cohort
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Started | 0 | 0 | 7 | 0 | 0
Completed | 0 | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: BAL101553 12 mg Cohort
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Started | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0
Period: BAL101553 15 mg Cohort
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Started | 0 | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort | Total
Number analyzed (Participants) | 5 | 5 | 7 | 5 | 4 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5 | 2 | 2 | 14
  >=65 years | 2 | 3 | 2 | 3 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.57) | 67.6 (6.27) | 57.7 (11.22) | 62.6 (12.10) | 57.8 (13.40) | 60.7 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 3 | 2 | 15
  Male | 1 | 3 | 3 | 2 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 3 | 6 | 5 | 4 | 23
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 5 | 5 | 6 | 4 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 7 | 5 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-Limiting Toxicities (DLTs) for Each Maximal Tolerated Dose (MTD)-Determining Dose Cohort
Description: A DLT was defined as a clinically-significant adverse event (AE) or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications. Any DLT had to be a toxicity considered at least possibly related to BAL101553 or the combination of BAL101553 and radiation.
Time Frame: Up to 10 weeks
Population: MTD-determining population: All patients who met any of the following criteria:
  * Received at least one dose of BAL101553 and has experienced a DLT;
  * Received ≥80% of their expected dose of BAL101553 and completed 6 weeks of combined treatment and 4 weeks of rest.
Measure: Number; unit: participants
Groups:
- BAL101553 4 mg MTD-determining Cohort: BAL101553 was given as an 4 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 6 mg MTD-determining Cohort: BAL101553 was given as an 6 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 8 mg MTD-determining Cohort: BAL101553 was given as an 8 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 12 mg MTD-determining Cohort: BAL101553 was given as an 12 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
- BAL101553 15 mg MTD-determining Cohort: BAL101553 was given as an 15 mg oral dose once daily (7 days per week) for 6 weeks, in combination with standard radiotherapy (RT)
Arm/Group | BAL101553 4 mg MTD-determining Cohort | BAL101553 6 mg MTD-determining Cohort | BAL101553 8 mg MTD-determining Cohort | BAL101553 12 mg MTD-determining Cohort | BAL101553 15 mg MTD-determining Cohort
Number analyzed (Participants) | 5 | 5 | 6 | 4 | 4
participants | 0 | 0 | 1 | 1 | 0

2. Secondary Outcome: Number of Patients With Grade 3 to Grade 5 Adverse Events (AEs)
Description: Common Terminology Criteria for Adverse Events (CTCAE) displayed by increasing severity grades 3 to 5 (CTCAE grade 3/4/5 )
Time Frame: up to 10 weeks
Population: All patients who received at least one full or partial dose of BAL101553 and had at least one post-baseline safety assessment was included in the safety analysis populations.
Measure: Count of Participants; unit: Participants
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
Number analyzed (Participants) | 5 | 5 | 7 | 5 | 4
Participants
  Number of patients with only unrelated CTCAE Grade 3/4/5 AEs | 1 | 2 | 1 | 2 | 1
  Number of patients with related CTCAE Grade 3/4/5 AEs | 1 | 1 | 1 | 1 | 0
  Number of patients without CTCAE Grade 3/4/5 AEs | 3 | 2 | 5 | 2 | 3

3. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time from Day 1 dosing to the date of death. Patients who have not died at study closure were censored at the time of last known alive.
Time Frame: Day 1 to date of death - up to 1679 days (4.6 years)
Population: Full analysis population (FAP) included all patients who received at least one partial or complete dose of study drug, based on the intent-to-treat principle. In this study the FAP corresponded to the safety population.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- All BAL101553 Treated Patients: OS is determined by Kaplan-Meier method for the safety population overall only, as predefined in the SAP. Due to the small number of patients, it is not possible to determine meaningfully comparable statistical values for the individual dose cohorts.
Arm/Group | All BAL101553 Treated Patients
Number analyzed (Participants) | 26
Days | 383.0 [273.0 to 552.0]

4. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS was the interval between Day 1 dosing and the earliest date of progression. Progression was defined as: an increase in tumor size of more than 25% or the appearance of new lesions on MRI scans, significant clinical deterioration not attributable to causes other than the tumor, or death from any cause.
  Patients who have not progressed or died at study closure were censored at the time of their last assessment without progression.
Time Frame: Day 1 to date of disease progression - 1092 days (3.0 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- All BAL101553 Treated Patients: PFS is determined by Kaplan-Meier method for the safety population overall only, as predefined in the SAP. Due to the small number of patients, it is not possible to determine meaningfully comparable statistical values for the individual dose cohorts.
Arm/Group | All BAL101553 Treated Patients
Number analyzed (Participants) | 26
Days | 247.0 [128.0 to 366.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 10 weeks from start of treatment, All-cause Mortality monitored up to 1679 days (4.6 years)
Description: Treatment-emergent events (TEAEs) were defined as all events occurring after BAL101553 treatment began
Arm/Group | BAL101553 4 mg Cohort | BAL101553 6 mg Cohort | BAL101553 8 mg Cohort | BAL101553 12 mg Cohort | BAL101553 15 mg Cohort
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/5 | 4/7 | 4/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/5 | 2/7 | 2/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 7/7 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAL101553 4 mg Cohort (N=5) | BAL101553 6 mg Cohort (N=5) | BAL101553 8 mg Cohort (N=7) | BAL101553 12 mg Cohort (N=5) | BAL101553 15 mg Cohort (N=4)
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAL101553 4 mg Cohort (N=5) | BAL101553 6 mg Cohort (N=5) | BAL101553 8 mg Cohort (N=7) | BAL101553 12 mg Cohort (N=5) | BAL101553 15 mg Cohort (N=4)
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood chloride decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0
Carbon dioxide increased (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0 | 1 | 2
Protein total decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 2 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 1 | 3
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Psychomotor skills impaired (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Slow speech (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Upper motor neurone lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 3 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Depilation (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 2
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1 | 3 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 4 | 5 | 3 | 3
Gait inability (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 2 | 3 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03250299/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03250299/SAP_001.pdf